CLINICAL TRIAL: NCT03177863
Title: Expectancy as Alternative to Treatment for Cervical Intraepithelial Neoplasia Grade 2 Among Women 25 - 30 Years of Age. A Multicenter Clinical Study
Brief Title: Expectancy as Alternative to Treatment for Cervical Intraepithelial Neoplasia Grade 2 Among Women 25 - 30 Years of Age
Acronym: EXCIN2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Björn Strander, Senior researcher, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EX CIN 2 001
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: CIN2; Therapy
Keywords: neoplasm; uterine cervix
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study cohort (Experimental): Healthy women 25 - 30 years of age with CIN2 who consent to inclusion and with no former history of CIN (any grade). The "intervention" is expectancy with clinical visits every 6 months. Women will leave study cohort if found with total regression (no CIN) or CIN3
  Interventions: Procedure: Expectancy

INTERVENTIONS:
Procedure: Expectancy — Clinical monitoring. See arm description

SUMMARY:
In the Swedish organised cervical screening program precursors of cervical cancer are detected and treated. Most precursor lesions detected by screening heal spontaneously. Those who progress do it slowly. There are three levels from light; CIN1, moderate; CIN2 to severe; CIN3. Women with CIN3 are always treated, regardless of age, according to current clinical guidelines. Women with CIN2 who are below the age of 25 years are offered active expectance for up to two years because there is good evidence that they will spontaneously heal their lesions (regression) in 40-70% of the cases during that time.

Method of treatment is today an excisional procedure of the cervix most often by Large loop excision of the transformation zone (LLETZ/LEEP) Treatment increases the risk of premature birth in a future pregnancy. In 2015 about 1800 excisional procedures of the transformation zone of the cervix were performed in the Västra Götalands regionen (VGR) om Sweden. The average age of first-time mothers in Sweden is rising and in 2014 it was 29 years. Postponed childbearing raises the question whether it is possible to refrain from surgery even for the group of women over 25 years old, with proven CIN2. Existing studies suggest that cure of CIN2 in the age group of and above 25 takes place in the same extent as under 25 years of age.There is lack of evidence concerning clinical follow-up.

In a prospective multicenter clinical cohort study (observational study) with careful monitoring, the investigators will examine what proportion of CIN2 changes regress spontaneously within two years in women, 25-30 years old, and if human papillomavirus (HPV) type 16 may can be a marker for poor regression in this group. Instead of LLETZ, active expectance is offered to women this age with CIN2 in five gynecological clinics in VGR. The study protocol includes gynecologist visits every 6 months for two years, including cytology, colposcopy and directed biopsies of the cervix. Power calculation shows 160 women needs to be included, which is expected to occur within one year from the start.

DETAILED DESCRIPTION:
Available in Swedish

ELIGIBILITY:
Inclusion Criteria:

* CIN 2
* Written consent

Exclusion Criteria:

* CIN (any grade) not resolved
* Former treatment of CIN
* Immunomodulating medication
* Pregnancy (at start of study)

Ages: 25 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Proportion of regress | 24 months from date of visit when CIN2 was diagnosed
  Proportion of women with CIN2 at inclusion who will regress to CIN1 or no evidence of disease

SECONDARY OUTCOMES:
Proportion of regress for women with HPV16 | Proportion of women with CIN2 at inclusion who will regress to CIN1 or no evidence of disease
  Proportion of women with CIN2 and HPV 16 at inclusion who will regress to CIN1 or no evidence of disease

CONTACTS AND LOCATIONS:
Overall Officials: Strander, Principal Investigator — Sahlgrenska Academy, Gothenburg University, Sweden
Locations (5):
- Sweden (5):
  - Södra Älvsborgs Sjukhus, Borås
  - Kungshöjds gynekologmottagning, Gothenburg
  - Frölunda specialistsjukhus, Gothenburg
  - Skaraborgs sjukhus, kvinnokliniken, Skövde
  - Norra Älvsborgs sjukhus, kvinnokliniken, Trollhättan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Massad LS, Einstein MH, Huh WK, Katki HA, Kinney WK, Schiffman M, Solomon D, Wentzensen N, Lawson HW; 2012 ASCCP Consensus Guidelines Conference. 2012 updated consensus guidelines for the management of abnormal cervical cancer screening tests and cancer precursors. Obstet Gynecol. 2013 Apr;121(4):829-846. doi: 10.1097/AOG.0b013e3182883a34. PMID 23635684
- [Background] Kyrgiou M, Mitra A, Arbyn M, Stasinou SM, Martin-Hirsch P, Bennett P, Paraskevaidis E. Fertility and early pregnancy outcomes after treatment for cervical intraepithelial neoplasia: systematic review and meta-analysis. BMJ. 2014 Oct 28;349:g6192. doi: 10.1136/bmj.g6192. PMID 25352501
- [Result] Wilkinson TM, Sykes PH, Simcock B, Petrich S. Recurrence of high-grade cervical abnormalities following conservative management of cervical intraepithelial neoplasia grade 2. Am J Obstet Gynecol. 2015 Jun;212(6):769.e1-7. doi: 10.1016/j.ajog.2015.01.010. Epub 2015 Jan 9. PMID 25582099
- [Result] Ostor AG. Natural history of cervical intraepithelial neoplasia: a critical review. Int J Gynecol Pathol. 1993 Apr;12(2):186-92. PMID 8463044
- [Result] Discacciati MG, de Souza CA, d'Otavianno MG, Angelo-Andrade LA, Westin MC, Rabelo-Santos SH, Zeferino LC. Outcome of expectant management of cervical intraepithelial neoplasia grade 2 in women followed for 12 months. Eur J Obstet Gynecol Reprod Biol. 2011 Apr;155(2):204-8. doi: 10.1016/j.ejogrb.2010.12.002. Epub 2010 Dec 28. PMID 21193261
- [Result] Guedes AC, Zeferino LC, Syrjanen KJ, Brenna SM. Short-term outcome of cervical intraepithelial neoplasia grade 2: considerations for management strategies and reproducibility of diagnosis. Anticancer Res. 2010 Jun;30(6):2319-23. PMID 20651386
- [Result] Ho GY, Einstein MH, Romney SL, Kadish AS, Abadi M, Mikhail M, Basu J, Thysen B, Reimers L, Palan PR, Trim S, Soroudi N, Burk RD; Albert Einstein Cervix Dysplasia Clinical Consortium. Risk factors for persistent cervical intraepithelial neoplasia grades 1 and 2: managed by watchful waiting. J Low Genit Tract Dis. 2011 Oct;15(4):268-75. doi: 10.1097/LGT.0b013e3182216fef. PMID 21811178
- [Result] Castle PE, Schiffman M, Wheeler CM, Solomon D. Evidence for frequent regression of cervical intraepithelial neoplasia-grade 2. Obstet Gynecol. 2009 Jan;113(1):18-25. doi: 10.1097/AOG.0b013e31818f5008. PMID 19104355